CLINICAL TRIAL: NCT01075490
Title: Neonatal Spinal Anesthesia: Effects of the Addition of Clonidine
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Alain Rochette, University Hospital of Montpellier
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UF7874
Record Dates: First submitted 2009-05-12; First posted 2010-02-25 (Estimated); Last update posted 2010-02-25 (Estimated); Status verified 2009-06

CONDITIONS: Spinal Anesthesia; Neonates
Keywords: spinal anesthesia; neonates; clonidine; post operative apnea
MeSH Terms: interventions — Clonidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- prematurely born, bupivacaine, placebo (Placebo Comparator)
  Interventions: Drug: clonidine
- prematurely born, bupivacaine, clonidine (Experimental)
  Interventions: Drug: clonidine
- term neonate, bupivacaine, placebo (Placebo Comparator)
  Interventions: Drug: clonidine
- term neonate, bupivacaine, clonidine (Experimental)
  Interventions: Drug: clonidine

INTERVENTIONS:
Drug: clonidine — addition of 1 µg/kg of clonidine to bupivacaine 1 mg/kg as spinal anesthesia
  Arms: prematurely born, bupivacaine, clonidine; term neonate, bupivacaine, clonidine
Drug: clonidine — equivalent volume of saline added to bupivacaine, 1 mg/kg as spinal anesthesia
  Arms: prematurely born, bupivacaine, placebo; term neonate, bupivacaine, placebo

SUMMARY:
This prospective, double blinded study investigates spinal anesthesia with or without clonidine added to bupivacaine in newborns. This study is based on duration measurement of spinal anesthesia and cardio respiratory recording during 24h for apnea detection.

DETAILED DESCRIPTION:
Ex premies and term neonates are two subgroups investigated separately. The overall objective is to validate lengthening of spinal anesthesia in newborns in order to avoid "rescue" general anesthesia that occur in 20-40 % of patients with plain bupivacaine.

ELIGIBILITY:
Inclusion Criteria:

* Newborns less than 60 weeks old post-conceptional, former premature or not
* Newborns requiring inguinal hernia or lower limbs surgery,
* infants needing no more critical care assistance
* Informed consent of parents

Exclusion Criteria:

* Spinal malformation,
* Coagulopathy,
* critical hemodynamics,
* uncontrolled neurologic or metabolic pathology.
* infection at injection point.

Max Age: 60 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2006-11; Primary Completion 2006-11 (Actual); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
number of "rescue" general anesthesia | end of surgery

SECONDARY OUTCOMES:
apnea and desaturation occurrence | during 24h
duration of spinal anesthesia | during 24h

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Capdevila, PhD, Study Chair — CHU de Montpellier, France; Alain Rochette, MD, Principal Investigator — CHU de Montpellier, France
Locations (1):
- CHU de Montpellier, Montpellier, France

REFERENCES:
- [Background] Rochette A, Raux O, Troncin R, Dadure C, Verdier R, Capdevila X. Clonidine prolongs spinal anesthesia in newborns: a prospective dose-ranging study. Anesth Analg. 2004 Jan;98(1):56-59. doi: 10.1213/01.ANE.0000093229.17729.6C. PMID 14693584
- [Background] Rochette A, Troncin R, Raux O, Dadure C, Lubrano JF, Barbotte E, Capdevila X. Clonidine added to bupivacaine in neonatal spinal anesthesia: a prospective comparison in 124 preterm and term infants. Paediatr Anaesth. 2005 Dec;15(12):1072-7. doi: 10.1111/j.1460-9592.2005.01664.x. PMID 16324026